CLINICAL TRIAL: NCT05922514
Title: Spontaneous Intracranial Hypotension Registry
Brief Title: A Clinical Registry of Spontaneous Intracranial Hypotension
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Waleed Brinjikji, Principal Investigator, Mayo Clinic
Other Study IDs: 21-006331
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Spontaneous Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 Baseline, 3 months, 1 year, 1.5 years, and 2 years Questionnaires: 170 participants with BERN imaging score with completion of baseline, 3 months, 1 year, 1.5 years, and 2 years questionnaires being : headache impact test (HIT-6), migraine disability assessment test (MIDAS), pain numerical rating scale (NRS), and spontaneous intracranial hypotension symptom severity scale (SIHSS).
  Each participant will keep a daily headache diary for 90 days.
  Interventions: Procedure: Transvenous Embolization of Cerebrospinal Fluid-Venous Fistula
- Group 2 Baseline, 7 days and 3 month, 1 year, 1.5 years, and 2 years Questionnaires: 30 participants with BERN imaging score with completion of baseline, 7 days, 3 months, 1 year, 1.5 years, and 2 years questionnaires being : headache impact test (HIT-6), migraine disability assessment test (MIDAS), pain numerical rating scale (NRS), and spontaneous intracranial hypotension symptom severity scale (SIHSS).
  Each participant will keep a daily headache diary for 90 days.
  Interventions: Procedure: Transvenous Embolization of Cerebrospinal Fluid-Venous Fistula

INTERVENTIONS:
Procedure: Transvenous Embolization of Cerebrospinal Fluid-Venous Fistula — Transvenous embolization of a cerebrospinal fluid-venous fistula performed via percutaneous venous access under fluoroscopic guidance. The procedure involves catheterization of the paraspinal or epidural venous system draining the fistula and delivery of an embolic agent to occlude the pathological venous outflow and eliminate CSF egress. The goal is to achieve durable fistula occlusion and resolution of spontaneous intracranial hypotension symptoms.

SUMMARY:
The purpose of this research is to determine the efficacy of paraspinal vein embolization for treatment of digital subtraction myelography (DSM) or CT myelography (CTM) confirmed cerebrospinal fluid (CSF)-venous fistulas so that researchers can inform the development and design of future clinical trials of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be patients who meet the International Classification of Headache - Disorders 3rd Edition (ICHD-3) criteria for a diagnosis of SIH or the Schievink criteria with imaging confirmed CSF-venous fistulas on DSM or CTM.
* Availability of a clinically prescribed contrast enhanced MRI positive for SIH.
* Negative urine or serum pregnancy test at time of study consent and three-months.

Exclusion Criteria:

* Patients who have a contraindication or inability to undergo the procedure (i.e., severe contrast allergy).
* Inability to provide informed consent.
* Expected inability to complete the follow-up assessment.
* Current pregnancy or breast-feeding during study enrollment (from consent to study conclusion approximately 90-days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being seen at Mayo Clinic in Rochester, Minnesota, for spontaneous intracranial hypotension (SIH) treatment evaluation by a neurologist with expertise in SIH. Patients would then be scheduled to meet with vascular radiology interventionalist for treatment (discussion and treatment(s) planning/scheduling purposes per standard of care. Patients would then speak with the study's coordinator to see if they would be interested to participant with and enroll in this study prior to SIH treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Impact Test (HIT-6) | Baseline, 3 months, 1 year, 1.5 years, 2 years
  HIT-6 is a 6-item validated headache assessment tool designed to provide a global measure of headache impact in social functioning, role functioning, vitality, cognition, psychological distress, and severity of headache. Total score ranges 36-78: 36-49: little or no impact; 50-55 some impact; 56-59 substantial impact; >60 severe impact.
Change in Bern SIH MRI Score | Baseline, 3 months, 1 year, 1.5 years, 2 years
  The Bern SIH MRI score is a validated 9-point score assessing the severity of imaging finding suggestive of SIH. Calculated by adding the individual components for a score range of 0-9. Classified as low, intermediate, or high probability of having a CSF leak based on total Bern SIH score of 2 points or fewer (low), 3-4 points (intermediate), or 5 points or more (high).

SECONDARY OUTCOMES:
Change in Pain Numerical Rating Scale (NRS) | Baseline, 3 months, 1 year, 1.5 years, 2 years
  Subjects are asked to rate pain intensity in the past 7 days using a scale of 0 is no pain and 10 is the worst imaginable pain.
Change in Migraine Disability Assessment (MIDAS) | Baseline, 3 months, 1 year, 1.5 years, 2 years
  MIDAS 5-item questionnaire to measure the impact of headaches on life. Subjects indicate how many days headaches have impacted a specific activity. Score ranges: 0-5: little or no disability; 6-10: mild disability; 11-20: moderate disability: 21+ severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Brinjikji, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials